CLINICAL TRIAL: NCT03782519
Title: Quality of Life of Frail Aged Patients in Incremental Hemodialysis: a Phase III Study
Brief Title: Quality of Life of Frail Aged Patients in Incremental Hemodialysis
Acronym: Qualifragilys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N/2016/75
Record Dates: First submitted 2018-12-07; First posted 2018-12-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Renal Dialysis; Kidney Failure, Chronic; Frailty
Keywords: Incremental Hemodialysis; Nephrology
MeSH Terms: conditions — Kidney Failure, Chronic; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental hemodialysis (Experimental): Patients who will begin HD with two treatment sessions per week
  Interventions: Other: Dialysis frequency reduction; Other: Frailty diagnosis
- Conventional hemodialysis (Active Comparator): Patients who will begin HD three times a week
  Interventions: Other: Frailty diagnosis

INTERVENTIONS:
Other: Dialysis frequency reduction — At initiation, frequency of dialysis will be reduced to 2 weekly sessions (incremental HD)
  Arms: Incremental hemodialysis
Other: Frailty diagnosis — Before randomization, we will determine whether patients are frail. We will define frailty as the presence of at least three of the following five conditions: malnourished according to dietitian assessment and/or short form of Mini Nutritional Assessment (MNA), grip strength and gait speed using participants' scores on the SF-36 Physical Functioning (PF) scale, exhaustion using in the quality of life questionnaire SF-36 vitality (VT) scale and physical activity according to patient assessment (one single question)

SUMMARY:
End stage renal disease (ESRD) is a major public health problem. The dialysis population is aging. As a result we observe a high prevalence of frailty among dialysis patients (ranges from 3 to 10 fold higher than in the comparably aged general public). Frailty is a medical syndrome characterized by diminished strength, endurance, and reduced physiologic function that increases an individual's vulnerability for developing increased dependency and/or death. Without systematic approach it is difficult for physicians to detect frailty phenotype which however might be reversible or attenuated by interventions. Fried et al. developed a frailty phenotype consisting of 3 or more of: unintentional weight loss, exhaustion, physical inactivity, slow gait speed, and weak grip strength. The primary care of hemodialysis patient is often supported by the nephrologist. Identification of frailty is integrated into the primary care setting as one of the steps necessary for the overall assessment of the person and planning to formal prevention interventions in an individualized care plan. Thrice-weekly hemodialysis (HD) schedules are the standard default hemodialysis prescription in Western countries, imposed in the 70s. For incremental HD, the weekly dose of dialysis is based on variety of clinical factors such as residual kidney function, volume status, cardiovascular symptoms, potassium level, nutritional status and, comorbid conditions. Incremental HD scheme generally starts with 2 weekly sessions and then periodic monitoring of criteria mentioned above are used to determine the timing for increasing dialysis dose and frequency to 3 weekly sessions.

An approach that integrates systematic frailty phenotype assessment by nephrologists and individualized incremental HD therapy can be beneficial within the first year of HD. It could optimize health-related quality of life and other pertinent outcomes without affecting negatively the quality of dialysis. The purpose of this study is to evaluate for frail aged incidents hemodialysis patients the impact of implementation of an incremental HD on HRQoL compared to conventional HD.

ELIGIBILITY:
Inclusion Criteria:

For all patients (incident HD patients):

* Patient aged over 60 years
* Signature of informed consent
* Affiliation to a French social security or receiving such a scheme
* Patient with Chronic Kidney Disease Stage 5 (GFR <15 ml/min/1.73m2)
* Urine output > 0,5 L per day
* Kru ≥ 2 ml/min
* Outpatient with scheduled start of HD
* Understand and read french

For randomized patients (frail incident HD patients):

- Frailty according to L. Fried criteria: score greater than or equal to 3/5

Exclusion Criteria:

* Inability to understand the reasons for the study; psychiatric disorders
* Active and/or treated neoplastic disease
* Scheduled kidney transplantation within 6 months
* Solid organ transplanted patient receiving immunosuppressive therapy
* Estimated life expectancy < 6 months
* Patient with diagnosis of severe chronic heart failure (> 2 congestive heart failure episodes requiring hospitalization in the year preceding the start of HD)
* Legal disability or limited legal capacity
* Patient without health insurance
* Pregnant
* Patient in the period of exclusion of another study
* Uncooperative patient

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 783 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Mental and physical health summary scores of the Medical Outcome Study - Short Form 36 (MOS SF-36) | One year after the initiation of HD
Symptom/problem, effects of kidney disease and burden of kidney disease dimensions of the Kidney Disease Quality of Life (KDQOL) | One year after the initiation of HD

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Courivaud, MD, PhD, Principal Investigator — Nephrology, Dialysis and Renal Transplantation - CHU Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiteni F, Pam A, Anota A, Vernerey D, Paget-Bailly S, Westeel V, Bonnetain F. Health-related quality-of-life as co-primary endpoint in randomized clinical trials in oncology. Expert Rev Anticancer Ther. 2015;15(8):885-91. doi: 10.1586/14737140.2015.1047768. Epub 2015 May 31. PMID 26027598